CLINICAL TRIAL: NCT06891508
Title: The Placenta-derived Secretome of Mesenchymal Stromal Cells as a Therapeutic Tool to Prevent Inflammation-induced Preterm Birth
Brief Title: The Placental Secretome as a Therapeutic Tool to Prevent Inflammation-induced Preterm Birth
Acronym: PLACENTOMICS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 7273
Record Dates: First submitted 2025-03-11; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Blood Specimen Collection; Cordocentesis

STUDY DESIGN:
Intervention Model Description: This study is interventional because of maternal peripheral blood sampling
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Women with spontaneous preterm birth (Experimental): Women enrolled in this study will undergo a venous blood draw (3 mL) via venipuncture from the antecubital fossa at the time of delivery. The placenta and amniochorionic membranes (hAM) will be collected within 30 minutes after delivery, performed via cesarean section. Additionally, a 3 mL sample of umbilical cord blood will be drawn from the residual cord attached to the placenta immediately after clamping.
  Interventions: Other: Venous blood sampling; Other: Tissues sampling; Other: Umbilical cord blood sampling
- Women with medically induced preterm birth (Active Comparator): Women enrolled in this study will undergo a venous blood draw (3 mL) via venipuncture from the antecubital fossa at the time of delivery. The placenta and amniochorionic membranes (hAM) will be collected within 30 minutes after delivery, performed via cesarean section. Additionally, a 3 mL sample of umbilical cord blood will be drawn from the residual cord attached to the placenta immediately after clamping.
  Interventions: Other: Venous blood sampling; Other: Tissues sampling; Other: Umbilical cord blood sampling
- Healthy women with at least two previous uncomplicated pregnancies (Active Comparator): Women enrolled in this study will undergo a venous blood draw (3 mL) via venipuncture from the antecubital fossa at the time of delivery. The placenta and amniochorionic membranes (hAM) will be collected within 30 minutes after delivery, performed via cesarean section. Additionally, a 3 mL sample of umbilical cord blood will be drawn from the residual cord attached to the placenta immediately after clamping.
  Interventions: Other: Venous blood sampling; Other: Tissues sampling; Other: Umbilical cord blood sampling

INTERVENTIONS:
Other: Venous blood sampling — Venous blood sampling (3 mL) via venipuncture from the antecubital fossa at the time of delivery
Other: Tissues sampling — Sampling of the placenta and amniochorionic membranes (hAM) at delivery
Other: Umbilical cord blood sampling — Umbilical cord blood sampling from the residual cord attached to the placenta immediately after clamping.

SUMMARY:
Preterm birth complicates 10% of all pregnancies and is the leading cause of perinatal morbidity and mortality worldwide. Intra-amniotic inflammation (IAI) and chorioamnionitis are well-established causes of PTB; however, a treatable infectious trigger is identified in only 50% of cases.In sterile IAI and/or preterm premature rupture of membranes (pPROM), there are currently no effective therapeutic options to reduce inflammation, promote amniotic sac healing, and prevent preterm birth. Growing evidence suggests that the secretome of mesenchymal stem cells (MSC) exhibits immunomodulatory and tissue-regenerative properties, making it a promising therapeutic tool for inflammatory disorders. Specifically, the conditioned medium from human amniotic mesenchymal stromal cells (CM-hAMSC) has been successfully used to treat various preclinical inflammatory disease models.

The aims of this study will be:1) to evaluate the activation of the NLRP3 inflammasome in hAM cells and peripheral blood mononuclear cells (PBMCs) from women with PTB. 2)To investigate the effect of CM-hAMSC on NLRP3 activation induced by lipopolysaccharide (LPS) and nigericin in cultured human amniotic epithelial cells (hAECs), amniotic mesenchymal stromal cells (hAMSCs), and PBMCs.

DETAILED DESCRIPTION:
Preterm birth complicates 10% of all pregnancies and is the leading cause of perinatal morbidity and mortality worldwide. Among all PTB cases, 70% occur spontaneously (SPTB), while the remaining 30% are medically indicated due to severe intrauterine growth restriction (IUGR). Intra-amniotic inflammation (IAI) and chorioamnionitis are well-established causes of SPTB; however, a treatable infectious trigger is identified in only 50% of cases.In sterile IAI and/or preterm premature rupture of membranes (pPROM), there are currently no effective therapeutic options to reduce inflammation, promote amniotic sac healing, and prevent preterm birth.Recent studies have identified the activation of the NLRP3 inflammasome in human amniotic membranes (hAM) as a key mechanism in the pathogenesis of SPTB. Targeting NLRP3 as a therapeutic approach for inflammatory diseases is rapidly advancing. Growing evidence suggests that the secretome of mesenchymal stem cells (MSC) exhibits immunomodulatory and tissue-regenerative properties, making it a promising therapeutic tool for inflammatory disorders. Specifically, the conditioned medium from human amniotic mesenchymal stromal cells (CM-hAMSC) has been successfully used to treat various preclinical inflammatory disease models.

The aims of this study will be:1) to evaluate the activation of the NLRP3 inflammasome in hAM cells and peripheral blood mononuclear cells (PBMCs) from women with PTB. 2)To investigate the effect of CM-hAMSC on NLRP3 activation induced by lipopolysaccharide (LPS) and nigericin in cultured human amniotic epithelial cells (hAECs), amniotic mesenchymal stromal cells (hAMSCs), and PBMCs.

ELIGIBILITY:
Inclusion Criteria:

* Full-term uncomplicated pregnancy, without any medical conditions or ongoing pharmacological treatment (control group).
* Pregnancy complicated by spontaneous preterm birth (gestational age 24-32 weeks).
* Pregnancy complicated by medically indicated preterm birth (gestational age 24-32 weeks).

Exclusion Criteria:

* Age <18 years
* Chronic infections (HIV or HCV)
* Cancer
* Multiple pregnancy
* Inability to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2028-03-20 (Estimated)

PRIMARY OUTCOMES:
Anti-inflammatory effects of conditioned medium | Through study completion, an average of 1 year
  To investigate the effect of CM-hAMSC on NLRP3 activation induced by lipopolysaccharide (LPS) and nigericin in cultured hAECs, hAMSCs, and PBMCs

SECONDARY OUTCOMES:
Inflammasome activation | Through study completion, an average of 1 year
  To assess NLRP3 inflammasome activation in hAM cells and peripheral blood mononuclear cells (PBMCs) from women with term or preterm birth, whether spontaneous or medically indicated.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Tersigni, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Ostetricia e Patologia Ostetrica, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No